CLINICAL TRIAL: NCT04514315
Title: Comparison of Outcomes for Minimally Invasive and Conventional Cardiac Valvular Surgery: A Prospective Cohort Study
Brief Title: Valvular Surgery: Minimally Invasive vs Conventional Sternotomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, William Kent, Dr. William Kent, University of Calgary
Other Study IDs: REB20-0859
Record Dates: First submitted 2020-07-15; First posted 2020-08-14 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Minimally Invasive Cardiac Valvular Surgery
Keywords: Minimally Invasive Valvular Surgery; Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Minimally invasive aortic valve surgery: Patients undergoing minimally invasive aortic valve surgery
  Interventions: Procedure: Minimally invasive cardiac valvular surgery
- Minimally invasive mitral valve surgery: Patients undergoing minimally invasive mitral valve surgery
  Interventions: Procedure: Minimally invasive cardiac valvular surgery
- Conventional aortic valve surgery: Patients undergoing conventional aortic valve surgery
  Interventions: Procedure: Conventional cardiac valvular surgery

INTERVENTIONS:
Procedure: Minimally invasive cardiac valvular surgery — Minimally invasive valve surgery via right mini-thoracotomy.
  Groups: Minimally invasive aortic valve surgery; Minimally invasive mitral valve surgery
Procedure: Conventional cardiac valvular surgery — Conventional valve surgery via full median sternotomy
  Groups: Conventional aortic valve surgery

SUMMARY:
The conventional approach to heart valve operations is through a sternotomy. This involves a vertical incision in the sternum (breastbone) to gain access to the heart and its related structures. Post-operative recovery after sternotomy can take anywhere from 6 weeks to 3 months due to the time required for the sternum to fully heal.

Minimally invasive valve surgery is a less invasive alternative to conventional open-heart surgery. At the Foothills Medical Centre, surgeons perform minimally invasive valve surgery through a technique called right mini-thoracotomy. This involves a small incision on the right upper chest and leaves the sternum fully intact. It is unclear whether minimally invasive valve surgery provides better clinical outcomes and quality of life compared to conventional open heart surgery.

The purpose of this research study is to compare the clinical outcomes of minimally invasive valve surgery via right mini-thoracotomy to conventional surgery via open-heart surgery. The results of this study will inform surgeons of the benefits and disadvantages of minimally invasive surgery compared to the current standards. This will help in developing better treatment strategies for patients requiring valve therapy.

DETAILED DESCRIPTION:
BACKGROUND & RATIONALE: The conventional approach to heart valve operations is open-heart surgery. This involves a vertical incision along the sternum (breastbone) and splitting it in half to gain access to the heart and its related structures. Open-heart surgery provides maximal exposure of the heart to the surgeon and results in good clinical outcome. However, post-operative recovery after open-heart surgery can take anywhere from 6 weeks to 3 months due to the time required for the sternum to fully heal. During this time patients can experience considerable pain and reduced mobility which have a significant negative impact on quality of life and productivity. Patients are also prone to major sternal complications such as wound opening and sternal infection, all of which may compromise respiratory function and overall recovery.

Minimally invasive valve surgery is a less invasive alternative to open-heart surgery. At the Foothills Medical Centre, surgeons perform minimally invasive valve surgery through a technique called right mini-thoracotomy. This involves a small incision on the right upper chest and leaves the sternum fully intact. This approach has been increasingly favoured and adopted by patients and physicians due to the benefits of avoiding sternal complications associated with open-heart surgery as well as cosmetic benefits. Despite these benefits, it is still unclear whether minimally invasive valve surgery provides better clinical outcomes and quality of life compared to conventional open-heart surgery.

RESEARCH QUESTION & OBJECTIVES: The aim of this observational research study is to assess the post-operative functional recovery and clinical outcomes of minimally invasive valve surgery via right mini-thoracotomy and conventional surgery via full median sternotomy. The objectives of this study are:

1. To assess post-operative functional recovery in minimally invasive and conventional valve surgery patients by assessing recovery of respiratory function, pain, physical function, and quality of life back to baseline.
2. To assess post-operative complications in minimally invasive and conventional valve surgery patients by assessing the incidence of early mortality, stroke, post-operative atrial fibrillation, permanent pacemaker implantation, paravalvular leak, pulmonary complication, wound infection, acute kidney injury, and reoperation.
3. To assess post-operative valve function in minimally invasive and conventional valve surgery patients by assessing valve gradients and degree of leakage.
4. To assess perioperative support for minimally invasive and conventional valve surgery patients by assessing ventilation time, cardiopulmonary bypass time, cross-clamp time, amount of blood transfusion, analgesic requirements, and length of ICU and hospital stay.

METHODS: The proposed clinical study is a single-center, prospective cohort study. All participants will undergo data collection procedures over a 12-month follow-up period. Specifically, data regarding demographics, medical history, and medications will be collected, and spirometry testing with a hand-held spirometer will be performed at baseline. Patients will be evaluated in hospital on post-op Day 3 and at discharge for pain, analgesic/antibiotic use, wound healing, any clinical events, quality of life (EQ-5D), and spirometry. Subsequently, patients will return to hospital for follow-up visits post operatively for physical examination, interview, additional quality of life questionnaires (EQ-5D, KCCQ-23, Health Assessment Questionnaire), and spirometry testing at 2 weeks, 6 weeks, and 3 months after surgery, with a final phone interview at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years of age
* Undergoing non-emergent isolated aortic valve or mitral valve surgery
* Full median sternotomy approach or minimally invasive approach via right anterior/anterolateral mini-thoracotomy
* English speaking
* Geographically accessible; able and willing to attend follow-up visits
* Written informed consent

Exclusion Criteria:

* Recent CPR
* Previous cardiac surgery
* Emergency surgery (operative intervention within 24 hours of assessment)
* Previous permanent pacemaker implantation
* Poor respiratory function - two or more measurements of FVC, FEV1, or PEF <80% of predicted value based on age, gender, and height at baseline
* History of a bleeding disorder
* Excessively poor baseline health-related quality of life or physical functioning that would preclude a reasonable expected post-operative recovery to baseline
* Active significant systemic infection, (e.g. endocarditis, sepsis) a history of recurrent systemic infections; or have taken an antibiotic within 2 weeks prior to surgery
* Cognitive impairment (e.g., confusion, dementia, Alzheimer's disease, current substance abuse) that would preclude completion of survey questions or following instructions to complete pulmonary function testing
* History of malignancy within the past year (except for squamous or basal cell carcinoma of the skin that has been treated, with no evidence of recurrence)
* Recent history of significant drug or alcohol abuse
* Participation in another study that would affect the ability to obtain adequate follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving a heart valve operation through either a minimally invasive approach via right mini-thoracotomy or conventional open-heart surgery via full median sternotomy at the Calgary Foothills Medical Centre.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Post-operative recovery of respiratory function (FVC) | 12 months
  Rate of post-operative recovery of respiratory function to baseline as measured by forced vital capacity (FVC) in litres from baseline to 12 months post-surgery. This measurement will be obtained by performing a pulmonary function testing (PFT) using a hand-held electronic spirometer.
Post-operative recovery of respiratory function (FEV1) | 12 months
  Rate of post-operative recovery of respiratory function to baseline as measured by forced expiratory volume (FEV1) in litres from baseline to 12 months post-surgery. This measurement will be obtained by performing a pulmonary function testing (PFT) using a hand-held electronic spirometer.
Post-operative recovery of respiratory function (PEF) | 12 months
  Rate of post-operative recovery of respiratory function to baseline as measured by peak expiratory flow (PEF) in litres/minute from baseline to 12 months post-surgery. This measurement will be obtained by performing a pulmonary function testing (PFT) using a hand-held electronic spirometer.
Post-operative pain | 12 months
  Severity of post-operative pain from baseline to 12 months post-surgery. Pain will be measured using an 11-point numeric rating scale (0 to 10). The scales will be associated with descriptors 0=none, 10=worst. Patients will be assessed for pain at the surgical incision sites (ie. sternum/rib/groin), chest, breast, neck, back, arms, and legs - areas of the body which may be affected by sternotomy or minimally invasive surgery. As pain might also interfere with function and mobility, participants will be asked to what degree the pain associated with their surgical incisions interfere with their ability to breath, cough, walk, and sleep.
Post-operative analgesic use | 12 months
  Type (narcotics vs non-narcotics) and amount of analgesic use in milligrams will be collected from baseline to 12 months post-surgery as indicators of pain.
Post-operative recovery of health-related quality of life (EQ5D) | 12 months
  Rate of post-operative recovery of health-related quality of life (HRQL) as determined by EQ5D questionnaire from baseline to 12 months post-surgery. The EQ-5D is a validated questionnaire which consists of two components: a self-reported measure of HRQL and a valuation of health states relative to full-health. The health status description component measures HRQL according to a five dimensional classification system. The dimensions are mobility, self-care, usual activities, pain and mood. There are five levels in each dimension resulting in 3125 theoretically possible health states which can be converted to a single index score.
Post-operative recovery of health-related quality of life (EQ VAS) | 12 months
  Rate of post-operative recovery of health-related quality of life (HRQL) as determined by EQ VAS (visual analogue scale) from baseline to 12 months post-surgery. The EQ-5D is a validated questionnaire which consists of a component using a visual analogue scale to determine self-reported measures of HRQL. The self-reported measure involves rating one's own health on a scale of 0-100 using a visual analogue scale where 100 represents the best health one can imagine and 0 representing the worst health.
Post-operative recovery of health-related quality of life (KCCQ-12) | 12 months
  Rate of post-operative recovery of health-related quality of life (HRQL) as determined by KCCQ-12 from baseline to 12 months post-surgery. The Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) is a validated self-administered questionnaire that independently measures the patient's perception of their health status using 12 items. The KCCQ-12 quantifies 4 distinct domains: symptom frequency, physical function, social limitation, and quality of life, from which an overall summary score can be derived. Scores are generated from each domain and scaled from 0 to 100 - 0 denoting the worst and 100 the best possible status.
Post-operative recovery of health-related quality of life (HAQ) | 12 months
  Rate of post-operative recovery of health-related quality of life (HRQL) as determined by HAQ from baseline to 12 months post-surgery. The Health Assessment Questionnaire (HAQ) is a validated index used to identify difficulty in performing activities of daily living. Questions require that participants identify how much difficulty they have had managing a variety of activities of daily living such as: dressing & grooming, arising, eating, walking, hygiene, reach, grip, and activities. This questionnaire focuses on both fine and gross motor skills which are greatly affected in heart surgery patients due to post-operative pain and discomfort. The highest score (indicating the greatest disability) within each of the eight dimensions is used to calculate the 'disability index'.
Post-operative complications | 12 months
  Post-operative complications including: early mortality, stroke, post-operative atrial fibrillation, permanent pacemaker implantation, paravalvular leak, pulmonary complication, wound infection, acute kidney injury, and reoperation from baseline to 12 months post-surgery.
Post-operative valve function | 12 months
  Post-operative valve function as determined by valve gradients and degree of leakage from baseline to 12 months post-surgery.
Perioperative outcomes | Up to 12 months
  Perioperative outcomes including: postoperative ventilation time, cardiopulmonary bypass time, cross-clamp time, amount of blood transfusion, returns to operating room, and length of ICU and hospital stay from baseline to discharge from hospital.
Health services resource usage | 12 months
  Health services resource usage using the items examined for the perioperative outcomes (ie. ventilation time, length of ICU and hospital stay, etc…) as well as any additional health care services after discharge ie. visits to health care provider, home care services, hospital admissions, and emergency visits from baseline to 12 months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: William Kent, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No